## **Child Assent Form**

**NCT number: TBD** 

Date: August 1, 2024 (last reviewed by IRB; original approval March 18, 2022)



**Department of Occupational Therapy** 

## Hi!

My name is Dr. Kelle. I would like to play some new games with you. Your parents know I am asking you to play games. Your teachers also know I am here to play games with you. They all said it is ok! The games will help us learn about feelings and how to feel calm and happy. We will play with your friends. We will have fun and you can earn prizes!

Would you like to play with me? It's ok to say no or to say yes.

[Wait for child response. If do not respond, show below and say "If you don't want to say it, you can point to yes or no here"]:



[Researcher document response on spreadsheet]